CLINICAL TRIAL: NCT05186337
Title: Efficacy of Functional Remediation for Older-Age Patients With Bipolar Disorder (FROA-BD) as Adjuntive to Pharmacological Treatment Versus Treatment as Usual (TAU)
Brief Title: Functional Remediation for Older Adults With Bipolar Disorder
Acronym: FROA-BD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Consorcio Centro de Investigación Biomédica en Red (CIBER) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PI20/00060
Record Dates: First submitted 2021-12-15; First posted 2022-01-11 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2023-08

CONDITIONS: Bipolar Disorder
Keywords: older adults; bipolar disorder; functional remediation; cognition; functioning; interventions
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Functional Remediation for Older-Age Patients With Bipolar Disorder (FROA-BD)
  Interventions: Behavioral: FROA-BD programme
- Control (No Intervention): The control group (42 patients) will not receive any type of add-on psychotherapy.

INTERVENTIONS:
Behavioral: FROA-BD programme — The experimental group (n=42) will receive a 4-month intervention consisting of 32 sessions of treatment.
  Arms: Experimental

SUMMARY:
Bipolar Disorder (BD) is a chronic and severe mental illness characterized by the emergence of alternating mood episodes which range from extreme depression to manic states. Beyond affective episodes, there is consensus considering that cognitive and functional impairment are also core features in a substantial proportion of patients suffering from this mental condition, being both of them responsible of a negative impact on perceived quality of life (QoL). Despite, the association between cognitive performance, clinical and functioning outcomes in patients with BD has been largely explored among adult and middle-aged patients, there is a dearth of research about aging process among older adults with bipolar disoder (OABD) as well as in the design of tailored intervention targeting older individuals. Due to the longer life expectancy and subsequent aging of the world's population, is becoming increasingly common that people presenting with chronic health condition, including BD, survives longer. Currently, it has been estimated roughly the 25% of whole BD population is over 60 years old and it is expected that this percentage will increase up to 50% by 2030. Consequently, there is an urgent need not only to explore specific implication in clinical and neurocognitive course and to investigate symptom development throughout this vital stage elder-life phase, but also to design specific interventions aimed to cope with special needs in this specific population.

DETAILED DESCRIPTION:
Study design: This is a single-center, single-blind, randomized, controlled test-retest clinical study to evaluate the efficacy of the FROA-BD in a representative sample of patients with BD over 60 years old. This study will be carried out in the Bipolar and Depressive Disorders Unit at the Hospital Clinic of Barcelona, which takes part of the Spanish network Center for Biomedical Research in Mental Health (CIBERSAM0029. It will include two parallel arms (1:1) in order to assess the efficacy of a new psychological intervention as add-on therapy compared with treatment as usual to enhance functional outcome in OABD. This project has been approved by the Ethical Comittee of the Hospital Clinic of Barcelona and it will be carried up in accordance with the ethical principles of the Declaration of Helsinki and Good Clinical Practice in compliance with the data protection law in force and anonymization of the collected information.

Procedure All participants will be examined at baseline prior to inclusion in the study, using an extensive battery of questionnaires and tools aimed to assess main demographic, clinical, functioning, quality of life, well-being, and neurocognitive variables. Once the baseline assessment has been carried out, patients will be randomly allocated into the experimental group, which will receive the FROA-BD programme, or to the control group, which will be treated as usual (TAU). Four months later, when the intervention will be finished, all study participants will be assessed, especially on those areas that are supposed to be targeted by the FROA-BD programme (functional outcome as the main outcome, and neurocognitive performance, clinical symptoms, and quality of life and well-being as secondary outcomes), trying to avoid potential re-assessment learning effect by using alternative versions or tests. Finally, one year after inclusion (8 months after completion of the intervention), a complete assessment, mostly identical to which was used at baseline, will be performed (See Figure 1). In addition to the aforementioned assessment visits, all participants will also be followed up pharmacologically at the Bipolar and Depressive Disorder Unit of the Hospital Clinic of Barcelona, following the guidelines of good clinical practice. Research members involved in assessment will be blind to condition group (FROA-BD or TAU). Two clinical neuropsychologist (therapist and co-therapist) blind to baseline assessment results will conduct the FROA-BD intervention.

Data collection

1. Demographic, clinical variables and comorbidity A semi-structured clinical interview based on the SCID-5 will be administered to gather main demographic and clinical variables. The HDRS and the YMRS will be used to evaluate the presence of depressive and manic symptomatology, respectively. The Cumulative Illness Rating Scale-Geriatrics (CIRS-G) Spanish version will be administered in order to assess the presence of any somatic comorbid condition. Medical records will be also reviewed and considered.
2. Psychosocial functioning, quality of life and well-being Functional outcome will be assessed by the means of the FAST. This interviewer-administered brief scale, which comprises 24 items, was specifically designed to explore functional difficulties in psychiatric population among six specific functional domains (autonomy, occupational functioning, cognitive functioning, financial issues, interpersonal relationships and leisure time). Overall scores range from 0 to 72, being higher scores indicators of a worse functional impairment.

   Quality of life and well-being will be assessed using the Spanish version of the Short Form-36 Health Survey (SF-36) and the Spanish version of the World Health Organisation-Five Well-Being Index (WHO-5), respectively. The SF-36 is self-administered questionnaire which consists of 36 questions measuring eight separate dimensions related to quality of life (physical functioning, role limitation-physical, role limitation-emotional, vitality, mental health, social functioning, pain, and general health). Higher scores indicate better quality of life. WHO-5 is a self-administered short test consisting of 5 items rated on a 6-point scale assessing how the individual has been feeling over the last two weeks. Raw score ranges from 0 to 25. The higher scores the better perceived subjective well-being. In order to obtain the feedback from the patients, we also will consider the patient's satisfaction with the intervention through a self-applied instrument measured in likert scale (from 0 to 10) where the maximum score corresponds to completely satisfied.
3. Cognitive Reserve The Cognitive Reserve Assessment Scale in Health (CRASH) is an interviewer-administered, quick and easy-to-apply tool which was designed to evaluate cognitive reserve in psychiatric patients, especially in those suffering from severe mental conditions. This 23-item scale assess the three domains: education, occupation and intellectual and leisure activities, which are the main domains involved in cognitive reserve. This scale provides an overall score as well as a score for each assessed domain. The maximum score is 90. Higher scores indicate higher cognitive reserve.
4. Neuropsychological assessment In this study we will to assess cognitive performance both from the subjective and objective perspective. For gathering data regarding subjective cognitive complaints, we will use the Cognitive Complaints in Bipolar Disorder Rating Assessment (COBRA). This self-administered instrument consist of 16 items which are rated on a 4-point scale ((0) never; (1) sometimes; (2) frequently; (3) always). COBRA total score results is calculated by totaling all item scores and higher scores indicate a worse subjective cognitive performance.

For the objective assessment of neurocognitive function two different batteries of tests have been selected depending of time-point assessment:

(I) Extended battery: Overall cognition will be assessed by means of the Mini Mental Status Examination (MMSE) and the Spanish version of the Screen for Cognitive Impairment in Psychiatry (SCIP-S). Both of these brief scales were specifically designed for detecting cognitive deficits, being the latter specific for psychiatric population. The SCIP-S has three alternative forms as three different time-points of the study in order to avoid learning effect bias.

The estimated Intelligence quotient (IQ) will be calculated based on the results in the Vocabulary subtest from the Wechsler Adult Intelligence Scale (WAIS-III).

The Executive functions will be measured through the computerized Wisconsin Card Sorting Test (WSCT), the Stroop Color-Word Test (SCWT); the Phonemic (F-A-S) component of the Controlled Oral Word Association Test (COWAT) the copy of the Rey Osterrieth Complex Figure (ROCF) and the Trail Making Test-Part B (TMT-B).

Attention will be assessed by using the computerized version of the Continuous Performance Test (CPT-II) and the Trail Making Test-Part A (TMT-A).

The Working memory index (WM) will be calculated based on the performance in three subtest from the WAIS-III: Arithmetic, Digits, and Letter-Number sequencing.

The assessment of the Processing speed index will comprise two subtests of the WAIS-III: the Symbol Search and the Digit-symbol Coding subtests from the WAIS-III.

Verbal Learning and Memory performance will be evaluated through the California Verbal Learning Test (CVLT).

To examine visual memory The Rey Osterrieth Complex Figure-inmediate recall (ROCF) will be administered.

Language domain will be examined by means of the Boston Naming Test (BNT) and the Categorical (Animal Naming) component of the COWAT.

Visuoespatial domain will be assessed by the Juice Line Orientation (JLO). This battery will be administered at baseline visit (V0) and 12-month follow-up visit after inclusion (V2), with the exception of vocabulary subtest which only will be applied at baseline visit since it is a measure of estimated IQ.

(II) Brief cognitive battery: In order to avoid potential learning effects, we selected a brief cognitive battery consisting of the SCIP-S form 2, the SCWT, the TMT part A and B, the CPT-II, and the semantic and phonemic components of the COWAT. This brief battery of test will be administered at post-intervention visit (V1), four months after inclusion.

ELIGIBILITY:
Inclusion Criteria:

1. meeting diagnostic criteria according to Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) for bipolar disorder, either subtype I or II;
2. being aged over 60 years old;
3. being in full or partial remission Young Mania Rating Scale (YMRS) ≤ 10, Hamilton Depression Rating Scale (HDRS) ≤ 14) at the time of the inclusion and assessment;
4. presence of mild to moderate functional impairment as measured by the Functional Assessment Short Test (FAST) ≥ 11
5. providing written informed consent to participate.

Exclusion Criteria:

1. presenting an Intelligence Quotient (IQ) lower than 85;
2. having been received any kind of structured psychological intervention in the six previous months;
3. presence of central nervous system (CNS) condition, other than psychiatric, than may influence neurocognitive performance, (such as neurological diseases) or any physical condition that may hamper participation or correct assimilation of the contents of the intervention, (such as severe visual and/or hearing impairment);
4. presenting any other comorbid psychiatric condition except for sleep and/or anxiety disorders, and
5. having received electroconvulsive therapy in the prior six months.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2023-03-15 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
The primary outcome measure will be changes in functioning assessed by means of the FAST from baseline to endpoint, post-intervention | 15 days
  The scale is interviewer-administered, designed for the assessment of psychosocial functioning. The 24 items of the scale are divided among 6 specific areas of functioning: autonomy, occupational functioning, cognitive functioning, financial issues, interpersonal relationships and leisure time. Each individual item is scored from 0 to 3. The global score (0-72) is obtained when the scores of each item are added up. The higher the score, the more serious the difficulties.

CONTACTS AND LOCATIONS:
Overall Officials: Jose Sanchez-Moreno, Principal Investigator — Consorcio Centro de Investigación Biomédica en Red (CIBER)
Locations (1):
- Hospital Clinic of Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No